CLINICAL TRIAL: NCT05053074
Title: Nasal High Flow (NHF) Bei COPD - Effekte Auf Die Ventilation im Wachzustand
Brief Title: Nasal High Flow (NHF) in COPD - Effects on Ventilation in Wakefulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Prof DR med, Clinical Director, Institut für Pneumologie Hagen Ambrock eV
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NHFwake2020
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: COPD
Keywords: Nasal High Flow; PaCO2; Tidal Volume; Washout Effect
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHF - NHF/CO2 (Experimental): Patients with chronic respiratory failure are treated with nasal high flow during wakefulness. First with NHF (30l/min) alone, then NHF (30l/min) plus 1% CO2.
  Interventions: Device: Nasal High Flow (NHF)
- NHF/CO2 - NHF (Experimental): Patients with chronic respiratory failure are treated with nasal high flow during wakefulness. First with NHF (30l/min) plus 1% CO2 , then NHF (30l/min) alone.
  Interventions: Device: Nasal High Flow (NHF)

INTERVENTIONS:
Device: Nasal High Flow (NHF) — Patients with chronic respiratory failure are treated for 1 h with NHF therapy and with individual O2 supplementation during wakefulness.
  Other Names: AIRVO2

SUMMARY:
Controlled randomized crossover trial in patients with chronic obstructive respiratory disease (COPD), who are treated with Nasal High Flow (NHF) therapy during wakefulness with a small amount of CO2 added to the inhaled air to keep the patients' PaCO2 stable despite the washout effect. Aim of the study is to examine respiratory rate, tidal volume and work of breathing under NHF without the CO2 washout effect.

DETAILED DESCRIPTION:
In this controlled randomized crossover trial, 10 stable patients with chronic obstructive respiratory disease (COPD) are treated with Nasal High Flow (NHF) therapy during wakefulness. NHF treatment will inevitably result in increased upper airway washout and thus in a slight reduction of PaCO2 of approximately 2 mmHg. For compensation, a small amount of CO2 is added to the inhaled air during this experimental situation, which keeps the patients' PaCO2 stable. This will allow to examine the effects of NHF therapy on respiratory rate, tidal volume and work of breathing, that are not attributable to the CO2 washout effect.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized COPD patients GOLD (3 and 4) in stable phase after an acute exacerbation.
* Written informed consent is required for participation.

Exclusion Criteria:

* Acute respiratory failure with clinical instability or respiratory acidosis defined by pH<7.35
* Severe acute physical illness that does not allow the subject to participate in a clinical trial
* Unable to give consent
* Language, cognitive, or other impairments that may prevent independent completion of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Minute Ventilation | up to 1 hour
  Difference in respiratory minute volume under NHF versus NHF/CO2.

SECONDARY OUTCOMES:
Tidal Volume | up to 1 hour
  Difference in tidal volume (VT) under NHF versus NHF/CO2
Respiratory Rate | up to 1 hour
  Difference in respiratory rate under NHF versus NHF/CO2.
Transcutaneous pCO2 | up to 1 hour
  Difference in transcutaneous pCO2 under NHF versus NHF/CO2.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, Professor, Principal Investigator — Evang. Kliniken Essen-Mitte gGmbH
Locations (1):
- Evang. Kliniken Essen-Mitte gGmbH, Essen, North Rhine-Westphalia, Germany